CLINICAL TRIAL: NCT01381757
Title: Uitlity of MODS for the Diagnosis of MDR-TB and Second-Line Antituberculous Drug Susceptibility Testing in Mali
Brief Title: Utility of MODS for Diagnosis of MDR-TB and Second-Line Antituberculous Drug Susceptibility Testing in Mali
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911175; 11-I-N175
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-03-05

CONDITIONS: Tuberculosis, Pulmonary; Mycobacterium Tuberculous; Antitubercular Agents; Tuberculosis, Mulutidrug-Resistant; Extensively Drug-Resistant; Extensibely Drug-Resistant Tuberculosis
Keywords: Extensively Drug-Resistant Tuberculosis; First-Line Antituberculous Drugs; Second-Line Antituberculous Drugs; Middlebrook Culture; Agar Proportion Method
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis; Extensively Drug-Resistant Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

-Tuberculosis (TB) is an infection of the lungs caused by bacteria. In Mali, TB is diagnosed with a test that is fast and inexpensive but not always accurate. The purpose of this study is to test a new method for diagnosing TB, called the microscopic-observation drug-susceptibility (MODS) test. The MODS test takes 7 days to show results. The test also gives information on which drugs will work best in each case.

Objective:

-To test a new method for diagnosing tuberculosis called the microscopic observation drug susceptibility test.

Eligibility:

* Participants must be 12 years of age or older.
* They must have a diagnosis of TB from a sputum smear, or have symptoms of TB and an x-ray indicating that TB is present.

Design:

* Participants will take part in the study from 6 months to 21 months and be assigned to one of three groups, depending on what type of TB they have.
* At the first visit, researchers ask questions about general health and symptoms of TB. They check vital signs, draw blood, and ask for a sputum sample. The blood is used to check for HIV infection and for the number of CD4 cells, which measures the severity of the HIV infection.
* The 2-, 5-, and 6-month visits are similar to the first. Those who do not have multidrug-resistant (MDR) TB will end their participation after the 6-month visit. MDR TB is tuberculosis that has not responded to isoniazid and rifampicin. Participants with MDR TB will remain in the study for 21 months.
* No treatment is provided as part of this study.

DETAILED DESCRIPTION:
Approximately one-third of the world s population is infected with tuberculosis (TB), and over 1 million deaths occur annually worldwide because of it (1,2). Accurate diagnosis and TB drug susceptibility testing is necessary to treat the infection appropriately and bring this epidemic under control. Inappropriate treatment of TB, on the other hand, has led to the recent spread in multidrug-resistant TB (MDR-TB), estimated to affect over half of million people worldwide (2,4,5). Sputum smear microscopy, the diagnostic method commonly used in developing countries, is not as sensitive at detecting TB as culture-based techniques utilized in developed countries. Furthermore, drug-susceptibility testing is not routinely performed in resource-limited settings. Consequently, many individuals with TB in developing countries are treated with inadequate regimens, and MDR-TB continues to spread.

The microscopic-observation drug-sensitivity (MODS) assay has been recently developed for rapid diagnosis of TB and simultaneous detection of resistance to first-line TB medications in resource-limited settings (11). MODS has been shown to be as sensitive as traditional culturebased methods for the detection of TB, providing results for drug susceptibility testing that are highly concordant with standard techniques (10).

We propose to study the utility of the MODS assay for the diagnosis of TB in subjects who are sputum-smear positive or sputum-smear negative, and those with chronic TB. Susceptibility testing will be performed for first-line antituberculous drugs and, subsequently, second-line drugs, if subjects are found to have MDR-TB. The first primary objective is to calculate the sensitivity of detection of the MODS assay, compared with the Middlebrook culture method, in subjects suspected of having TB who are sputum-smear positive by microscopy. The second primary objective is to calculate the concordance of drug-susceptibility testing between the MODS assay and the agar proportion method for subjects who are sputum-smear positive, sputum-smear negative, or diagnosed with chronic TB.

Secondary objectives include evaluating the utility of the MODS assay in the diagnosis of TB in subjects who are sputum-smear negative and those with chronic TB, the performance of second-line drug-susceptibility testing using the MODS assay in subjects diagnosed with MDRTB, the utility of the MODS assay in the diagnosis of TB in subjects coinfected with human immunodeficiency virus (HIV)-1 or -2, and the ability of the MODS assay to identify nontuberculous mycobacteria in subjects harboring these organisms.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals (12 years of age) who meet the following criteria are eligible for enrollment in the study:

Have a sputum smear that is positive for acid-fast bacilli by microscopy or have clinical symptoms and abnormal findings compatible with active TB on a previously performed chest radiograph.

Have either completed at least 5 months of treatment with antituberculous therapy within the past year or have not received any antituberculous treatment in the preceding 5 years.

Willingness to provide a sputum sample for the study.

Ability to follow verbal instructions for producing sputum.

Willingness to undergo testing for HIV.

Willingness to allow storage of samples for future research.

EXCLUSION CRITERIA:

Subjects who meet any of the following criteria are not eligible for enrollment in the study:

Any condition that in the investigator s opinion places the subject at undue risk by participating in the study.

Subjects younger than 12 years of age will be excluded from the study due to the difficulty of obtaining adequate sputum samples for the diagnosis of TB in this population and because there are no means for obtaining gastric aspirates at the reference centers.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-05-31; Study Completion 2013-03-05

CONTACTS AND LOCATIONS:
Overall Officials: Sophia B Siddiqui, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- National Institute of Allergy and Infectious Diseases (NIAID), 9000 Rockville Pi, Bethesda, Maryland, United States
- University of Bamako, Bamako, Mali

REFERENCES:
- [Background] Chan ED, Iseman MD. Multidrug-resistant and extensively drug-resistant tuberculosis: a review. Curr Opin Infect Dis. 2008 Dec;21(6):587-95. doi: 10.1097/QCO.0b013e328319bce6. PMID 18978526
- [Background] Nathanson E, Nunn P, Uplekar M, Floyd K, Jaramillo E, Lonnroth K, Weil D, Raviglione M. MDR tuberculosis--critical steps for prevention and control. N Engl J Med. 2010 Sep 9;363(11):1050-8. doi: 10.1056/NEJMra0908076. No abstract available. PMID 20825317
- [Background] Gandhi NR, Nunn P, Dheda K, Schaaf HS, Zignol M, van Soolingen D, Jensen P, Bayona J. Multidrug-resistant and extensively drug-resistant tuberculosis: a threat to global control of tuberculosis. Lancet. 2010 May 22;375(9728):1830-43. doi: 10.1016/S0140-6736(10)60410-2. PMID 20488523